CLINICAL TRIAL: NCT06060587
Title: A Randomized Phase II Study of ADT + Abiraterone Versus ADT + Docetaxel + Abiraterone in Patients With Low Volume Metastatic Hormone Sensitive Prostate Cancer
Brief Title: Randomized Phase II Study of ADT + Abiraterone vs ADT + Docetaxel + Abiraterone
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left institution
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU 23U08; NCI-2023-07135 (Registry Identifier: CTRP); STU00220128 (Registry Identifier: Northwestern IRB); P30CA060553 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triplet Arm (Experimental): Abiraterone+Docetaxel+ADT
  Abiraterone Abiraterone acetate will be four (250 mg) tablets (total dose/day 1000 mg). Abiraterone administration is per a 12-week cycle.
  Abiraterone must be taken with prednisone. Prednisone will be provided as 5 mg tablets.
  Docetaxel Docetaxel on day 1 of each 21-day cycle, 75 mg/m2 via IV. Dexamethasone will be self-administered by the patient at 16 mg per day for 3 days starting 1 day prior to docetaxel infusion.
  ADT Patients may be started on an LHRH agonist or antagonist , the selection of the agent is left to the treating investigator for ADT.
  Interventions: Drug: Docetaxel; Drug: ADT; Drug: Abiraterone
- Doublet Arm (Active Comparator): Abiraterone+ADT
  Abiraterone Abiraterone acetate will be four (250 mg) tablets (total dose/day 1000 mg). Abiraterone administration is per a 12-week cycle.
  Treatment of abiraterone should start ≤14 days after patient randomization.
  Abiraterone must be taken with prednisone. Prednisone will be provided as 5 mg tablets.
  Docetaxel Docetaxel on day 1 of each 21-day cycle, 75 mg/m2 via IV. Prior to docetaxel, dexamethasone administration is recommended as discussed, but can be adjusted or altered per the treating investigator's discretion. Dexamethasone will be self-administered by the patient at 16 mg per day for 3 days starting 1 day prior to docetaxel infusion.
  Interventions: Drug: ADT; Drug: Abiraterone

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 via IV
  Arms: Triplet Arm
Drug: ADT — Prior to randomization as part of standard of care.
Drug: Abiraterone — 1000 mg by mouth

SUMMARY:
This is a phase II, randomized, open label study comparing first line therapy with AThis is a phase II, randomized, open label study comparing first line therapy with ADT + abiraterone (doublet arm) or ADT + abiraterone + docetaxel (triplet arm) in low volume, metastatic hormone sensitive prostate cancer (mHSPC).

This is a phase II, randomized, open label study comparing first line therapy with Androgen Deprivation Therapy (ADT) + abiraterone (doublet arm) or ADT + abiraterone + docetaxel (triplet arm) in low volume, metastatic hormone sensitive prostate cancer (mHSPC).

The hypothesis being asked in this trial is whether first line treatment with ADT plus an androgen receptor pathway inhibitor (abiraterone) as a doublet regimen compared to ADT plus an androgen receptor pathway inhibitor (abiraterone) and docetaxel, as a triplet regimen results in superior outcomes for patients with low volume mHSPC.

We plan to enroll patients with mHPSC that meet the CHAARTED criteria for low disease volume. Patients will be randomized 1:1 to either treatment arm:

* doublet arm: abiraterone +ADT or
* triplet arm: abiraterone + ADT + docetaxel.

All subjects must receive ADT of the Investigator's choice (LHRH agonist/antagonists or orchiectomy) as standard therapy, started = 12 weeks before randomization.

DETAILED DESCRIPTION:
Primary Objective:

1. To assess Progression Free Survival (PFS) for each treatment arms (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy

Secondary Objective:

1. To assess Overall Survival (OS) for each treatment arm (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy
2. To assess PSA Response Rate for each treatment arm (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy
3. To assess ORR with measurable disease at baseline for each treatment arm for (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy
4. Assessment of Time to castration resistant prostate cancer for each treatment arm (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy
5. Assess time to initiation of subsequent anti-neoplastic therapy for each treatment arm (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy

Exploratory Objectives:

1. Assess Quality of Life (QoL) via the FACT-P QoL assessment tool (Appendix A QoL Survey FACT-P) for each treatment arm (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy
2. Assessment of Rates of Adverse Events (AEs)/Serious adverse events (SAEs) for each treatment arm (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in safety

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed PCa and imaging evidence of metastatic disease on CT, MRI, and/or bone scan. A PSMA PET scan may be used, but findings confirming metastatic disease (ex. A lymph node > 1 cm or a bone lesion) must be observed on the CT portion of the scan.
* Patients must have low volume metastatic disease per the CHAARTED [1, 2] criteria; Low volume is defined as metastasis in lymph nodes outside of the pelvis and/or boney lesions (< 4 boney lesions, none outside of the axial skeleton). No visceral metastasis allowed. Metastatic disease must be documented either by a positive bone scan, contrast-enhanced abdominal/pelvic/chest computed tomography (CT) scan, magnetic resonance imaging scan or a prostate-specific membrane antigen (PSMA) PET scan. If a PSMA PET scan is used, the CT portion must confirm lymph node enlargement > 1cm or evidence of sclerosis for boney lesions. Metastatic disease is defined as either malignant lesions in the bone and/or measurable lymph nodes above the aortic bifurcation. Only patients with non-regional lymph node metastases (M1a) and/or bone metastases (M1B) will be eligible.
* Patients must have measurable disease as determined per RECIST version 1.1 See protocol for the evaluation of measurable disease. Lymph nodes are measurable if the short axis diameter is ≥ 10mm.
* Patient must be candidates for ADT, docetaxel and abiraterone therapy per treating investigator's judgment.
* Patients may have started ADT (LHRH agonist/antagonist or orchiectomy) for ≤ 12 weeks before randomization, with or without first generation anti-androgen.
* Patients must exhibit a/an ECOG performance status of ≤ 1.
* Patients must have adequate organ and bone marrow function as defined in the protocol.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* If a patient has known brain metastases, they must have received radiation per SOC to control disease to be eligible for this trial.
* The effects of abiraterone and docetaxel on the developing human fetus are unknown. For this reason and because chemotherapy agents as well as other therapeutic agents used in this trial are known to be teratogenic: patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) nor donate sperm, from time of informed consent, for the duration of study participation, and for 3 months following completion of abiraterone and 6 months following completion of docetaxel therapy. Should a patient's partner become pregnant or suspect they are pregnant while patient's partner is participating in this study, patient's partner should inform their treating physician immediately.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior treatment with:
* LHRH agonist/antagonist started > than 12 weeks before randomization NOTE: Use of androgen deprivation therapy (ADT) prior to the diagnosis of metastatic disease is allowed (see Inclusion Criteria 3.1.5 & Section 4 Treatment Plan for full information)
* Second generation ARPIs such as enzalutamide, ARN-509, abiraterone, other investigational AR inhibitors
* Cytochrome P17 enzyme inhibitors such as abiraterone acetate or oral ketoconazole as antineoplastic treatment for prostate cancer.
* Chemotherapy or immunotherapy for prostate cancer prior to randomization except as described in Inclusion criteria 3.1.5
* Treatment with radiotherapy (external beam radiation therapy, brachytherapy, or radiopharmaceuticals) within 2 weeks before randomization
* Previous (within 28 days before the start of study drug or 5 half-lives of the investigational treatment of the previous study, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s).
* Known hypersensitivity to any of the study drugs, study drug classes or excipients in the formation of any of the study drugs
* Contraindication to both CT and MRI contrast agent
* Had any of the following within 6 months before randomization: stroke, myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, congestive heart failure
* Uncontrolled hypertension as indicated by a resting systolic blood pressure (BP) ≥ 160 mmHg or diastolic BP ≥ 100 mmHg despite medical management
* Patients who are unable to swallow oral medication, have malabsorption syndrome, have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, small bowel resection) or any other uncontrolled gastrointestinal condition (e.g., nausea, diarrhea, or vomiting) that might impair the oral bioavailability of any of the study drugs
* Patients with history of or evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with history of or evidence of chronic hepatitis C virus (HCV) infection, must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) must have no detectable viral load on a stable antiviral regimen and have a CD4 count ≥ 200/mcL.
* Patients with chronic liver disease with a need for treatment
* Prior systemic treatment with an azole drug (e.g., fluconazole, itraconazole) within 4 weeks of randomization,
* Concomitant use of strong CYP3A4 inhibitors (see Appendix C)
* Patients who have an uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:
* Ongoing or active infection requiring systemic treatment
* Cardiac arrhythmia uncontrolled with medical management
* Any other illness or condition or clinical laboratory finding that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Major surgery within past 30 days
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* Any other serious or unstable illness, or medical, social, or psychological condition, that could jeopardize the safety of the subject and/or his/her compliance with study procedures, or may interfere with the subject's participation in the study or evaluation of the study results

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2030-12-22 (Estimated)

PRIMARY OUTCOMES:
Assess Progression Free Survival (PFS) | Up to 1 year after completion of study treatment
  Calculated the progression-free survival time as the time that elapses between the date of randomization and the day of first documented disease progression (per RECIST 1.1 or PCWG3) or death from any cause for all evaluable patients. PFS will be calculated based on the Kaplan-Meier estimates of PFS for each treatment arm (abiraterone+docetaxel+ADT compared to abiraterone+ADT).

SECONDARY OUTCOMES:
Assess Overall Survival (OS) | Up to 1 year after completion of study treatment
  To assess the OS, this is defined as the time from date of randomization until time to death from any cause for all evaluable patients. OS will be calculated based on the Kaplan-Meier estimates of OS.
Assess PSA Response Rate | 6 months (+/- 30 days) after randomization
  The PSA level drawn 6 months (+/- 30 days) after randomization will be used to assess PSA response.
Assessment of Time to castration resistant prostate cancer | Up to 1 year after completion of study treatment
  This endpoint will calculate the time to the development of castration resistance from date of randomization to the time of PSA progression with serum testosterone level being at ≤ 50 ng/ml
Assess time to compare for any difference in efficacy between arms | Up to 1 year after completion of study treatment
  This endpoint will calculate the time to the initiation of the subsequent anti-neoplastic therapy for each treatment arm from the date of randomization to the date of initiation of the next (non-study) anti-neoplastic agent for prostate cancer.

OTHER OUTCOMES:
Assess Quality of Life (QoL) | Time between the initiation of trial therapy to 30 days from the last dose of study drug
  FACT-P QoL assessment tool for each treatment arm (abiraterone+docetaxel+ADT and abiraterone+ADT) to compare for any difference in efficacy
Assessment of Rates of Adverse Events (AEs)/Serious adverse events (SAEs) | Time between the initiation of trial therapy to 30 days from the last dose of study drug
  To assess the rate of adverse events for each treatment arm. Safety will be measured as the frequency of AEs by type, severity (grade), timing and attribution to trial therapy (per NCI CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fenton, MD, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States